CLINICAL TRIAL: NCT05896904
Title: Clinical Comparison of Patients With Transthyretin Cardiac Amyloidosis and Patients With Heart Failure With Reduced Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Steen Hvitfeldt Poulsen, Professor, Aarhus University Hospital Skejby
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1-10-72-380-21
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Transthyretin Amyloid Cardiomyopathy; Heart Failure
Keywords: Heart Failure; Echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echocardiography (Experimental)
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography

SUMMARY:
Clinical comparison of patients with transthyretin cardiac amyloidosis and patients with heart failure with reduced ejection fraction

ELIGIBILITY:
Inclusion Criteria:

* Age >65
* ATTRwt diagnosis for patients, either with DPD-scintigraphy or myocardiac biopsy
* informed consent

Exclusion Criteria:

* Alder <65
* No ATTRwt diagnosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
intraventricular wall thickness | 1 year
  echocardiographic measurement

CONTACTS AND LOCATIONS:
Overall Officials: Valentin R Klarskov, Bachelor, Principal Investigator — Clinic of heart diseases, AUH.
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No